CLINICAL TRIAL: NCT01607671
Title: Can Urgent Reduction of Intraocular Pressure With Ophthalmic Timolol Improve Recovery From Non-arteritic Anterior Ischemic Optic Neuropathy (NAION): a Randomized Study.
Brief Title: Treatment Study for Ischemic Optic Neuropathy With Opthalmic Timolol Maleate 0.5%
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit participants from recruiting sites.
Sponsor: Fraser Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAION-001
Record Dates: First submitted 2012-05-25; First posted 2012-05-30 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Optic Neuropathy, Ischemic; Anterior Ischemic Optic Neuropathy; Ischemic Optic Neuropathy; Optic Neuropathy, Anterior Ischemic
Keywords: Ischemic; Optic Neuropathy; Non-Arteritic Anterior Ischemic Optic Neuropathy; NAION; Ischemic Optic Neuropathy; Intraocular Pressure
MeSH Terms: conditions — Optic Neuropathy, Ischemic; Ischemia; Optic Nerve Diseases | interventions — Timolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Timolol (Experimental): This group will receive ophthalmic Timolol maleate 0.5%, 1 drop to the effected eye twice daily for 4 weeks.
  Interventions: Drug: Timolol maleate
- Standard Care (No Intervention): This group will be treated with current standard care. This does not include Timolol or other medications to reduce intraocular pressure.

INTERVENTIONS:
Drug: Timolol maleate — Timolol 0.5% 1 drop twice daily to the effected eye for 4 weeks.
  Other Names: Timoptic.; Timolol.; Timolol maleate.
  Arms: Timolol

SUMMARY:
The purpose of this study is to evaluate the feasibility of rapid evaluation and administration of ophthalmic Timolol maleate in the treatment of non-arteritic anterior ischemic optic neuropathy. Secondary goals are to evaluate if such treatment reduces the progression or improves recovery of patients who are randomly assigned to treatment versus standard of care.

DETAILED DESCRIPTION:
Non-arteritic anterior ischemic optic neuropathy (NAION) currently has no widely accepted acute treatment to improve recovery or prevent progression in the first month. It causes monocular vision loss with potential second eye involvement in 15% at 5 years. This leads to significant disability. It is the most common acute optic neuropathy in patients over 55 years of age. The final mechanism of injury is believed to be ischemic. Increasing perfusion of the optic nerve may reduce damage and prevent progression. Reduction in intraocular pressure has been shown to increase optic disc perfusion in animal models. Timolol maleate is a widely used medication for Glaucoma that reduces intraocular pressure. Treatment with Timolol maleate may improve optic disc perfusion in NAION and reduce ischemic damage from this condition. This study aims to enroll and treat patients with Timolol maleate 0.5% within 48 hours of symptom onset to assess feasibility of the study design and potential benefit of rapid intraocular pressure reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age >40
* Sudden, painless monocular vision loss with edema of the optic disc
* Clinical diagnosis is Non-Arteritic Anterior Ischemic Optic Neuropathy
* Relative Afferent Pupil Defect (RAPD) at first study visit

Exclusion Criteria:

* Onset of vision loss >48 hours from time of enrollment
* History of Asthma or COPD
* History of Heart Block or Sinus Bradycardia
* Allergy to any beta blocker
* History of Multiple Sclerosis or optic neuropathy
* Active Ocular Inflammation on examination
* Currently being treated for Cancer or systemic vasculitis
* History of Glaucoma or use of medications that lower IOP
* Symptomatic cataract, retinopathy, macular disease or amblyopia in the symptomatic eye
* IOP of <10 at baseline
* Ocular surgery in past three months
* Women who are pregnant, breast-feeding or may become pregnant
* Inability to provide informed consent or follow up at three months
* Currently enrolled in any other study drug trial or previously enrolled in this study

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate of patients during the one year study to assess feasibility of a larger study | 12 months
  This is to define the feasabilty of the study design for a larger study.
Number of patients with adverse events | 12 months

SECONDARY OUTCOMES:
Change in visual acuity at enrollment and three month follow up using a logMAR scale. | Enrolment, Within 48 hours of enrollment , 1 month, 3 months.
  This will evaluate the change in visual acuity as a measure of visual function.
Change in the mean deviation of actual versus predicted sensitivity of the visual field. | 48 hours after enrollment, 1 month, 3 months
  Using a a Haag-Streit Octopus 900 with white on white TOP 30-2 visual field program, the mean deviation will be compared at various time points to assess for improving visual function as it relates to the field of vision.
Change in Colour vision as measured by HRR colour plates. | Within 48 hours of enrollment, 1 month, 3 months
  The total number of colour plates seen will be counted and compared to baseline as a measure of visual recovery as it effects colour vision.
Change in contrast sensitivity will be measured using the Pelli-Robson contrast sensitivity chart. | 48 hours from enrollment, 1 month, 3 months.
  The Pelli-Robson contrast sensitivity chart is another method to assess visual function. The change in total number of plates seen will be compared at the various time points.

CONTACTS AND LOCATIONS:
Overall Officials: Martin A SuttonBrown, MD, Principal Investigator — Fraser Health Region
Locations (1):
- Jim Pattison Outpatient Care and Surgery Centre, 3C Neurology, Surrey, British Columbia, Canada

REFERENCES:
- [Background] Atkins EJ, Bruce BB, Newman NJ, Biousse V. Treatment of nonarteritic anterior ischemic optic neuropathy. Surv Ophthalmol. 2010 Jan-Feb;55(1):47-63. doi: 10.1016/j.survophthal.2009.06.008. PMID 20006051
- [Background] Glucksberg MR, Dunn R. Direct measurement of retinal microvascular pressures in the live, anesthetized cat. Microvasc Res. 1993 Mar;45(2):158-65. doi: 10.1006/mvre.1993.1015. PMID 8361399
- [Background] Maepea O. Pressures in the anterior ciliary arteries, choroidal veins and choriocapillaris. Exp Eye Res. 1992 May;54(5):731-6. doi: 10.1016/0014-4835(92)90028-q. PMID 1623958
- [Background] Wilhelm B, Ludtke H, Wilhelm H; BRAION Study Group. Efficacy and tolerability of 0.2% brimonidine tartrate for the treatment of acute non-arteritic anterior ischemic optic neuropathy (NAION): a 3-month, double-masked, randomised, placebo-controlled trial. Graefes Arch Clin Exp Ophthalmol. 2006 May;244(5):551-8. doi: 10.1007/s00417-005-0102-8. Epub 2005 Sep 8. PMID 16151785
- [Background] Optic nerve decompression surgery for nonarteritic anterior ischemic optic neuropathy (NAION) is not effective and may be harmful. The Ischemic Optic Neuropathy Decompression Trial Research Group. JAMA. 1995 Feb 22;273(8):625-32. PMID 7844872